CLINICAL TRIAL: NCT00463424
Title: NeuFlex and Swanson Metacarpophalangeal Implants for Rheumatoid Arthritis: a Prospective Randomized Controlled Clinical Trial
Brief Title: Comparison of NeuFlex and Swanson Metacarpophalangeal Implants for Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: DePuy Orthopaedics (Industry); Stryker Trauma and Extremities (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB#2K-049C
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Metacarpophalangeal Joint; Arthroplasty, Replacement; Range of Motion, Articular; Randomized Controlled Trials; Swanson; NeuFlex
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NeuFlex metacarpophalangeal implant
Device: Swanson metacarpophalangeal implant

SUMMARY:
The main hypotheses for this study are as follows:

1. The use of NeuFlex implant results in flexion in the fourth and fifth MP joints that is at least 10 degrees greater than with teh use of the Swanson implant.
2. The use of the NeuFlex implant is associated with a significantly (2.5 kg or more) greater grip strength than with the use of the Swanson implant.

DETAILED DESCRIPTION:
Many studies have evaluated metacarpophalangeal joint (MP) range of motion following Swanson arthroplasty. These studies report that overall MP flexion is restricted postoperatively. They do not usually report individual range of motion values for each digit. Therefore one cannot identify if the degree of MP flexion restriction differs by digit.

We, and others, have observed that MP flexion is particularly restricted in the ring and litter finger following Swanson arthroplasty.

There is a new implant (NeuFlex), which instead of being introduced in full extension, like the Swanson implant, has a resting position of 30 degrees of flexion. As MP flexion is particularly restricted in the ring and little finger, an implant that by design encourages flexion may be helpful. A need exists to establish if the use of the NeuFlex implant produces greater MP flexion in the ring and little finger where restricted flexion has been identified as a problem.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis
* primary metacarpophalangeal arthroplasty of all 4 digits

Exclusion Criteria:

* diagnosis of other connective tissue disorder (e.g. SLE, MCTD)
* previous surgery of MP joints
* revision metacarpophalangeal arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2000-10; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Maximum active postoperative MP flexion

SECONDARY OUTCOMES:
Maximum active postoperative MP extension
Maximum active postoperative MP arc of motion
Ulnar drift
Jamar grip strength
Sollerman Hand Function Score
Michigan Hand Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Earl R Bogoch, MD, Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Delaney R, Trail IA, Nuttall D. A comparative study of outcome between the Neuflex and Swanson metacarpophalangeal joint replacements. J Hand Surg Br. 2005 Feb;30(1):3-7. doi: 10.1016/j.jhsb.2004.10.013. PMID 15620484
- [Background] Erdogan A, Weiss AP. [NeuFlex Silastic implant in metacarpophalangeal joint arthroplasty]. Orthopade. 2003 Sep;32(9):789-93. doi: 10.1007/s00132-003-0524-0. German. PMID 14508644
- [Background] Joyce TI, Unsworth A. NeuFlex metacarpophalangeal prostheses tested in vitro. Proc Inst Mech Eng H. 2005;219(2):105-10. doi: 10.1243/095441105X9192. PMID 15819481
- [Background] Weiss AP, Moore DC, Infantolino C, Crisco JJ, Akelman E, McGovern RD. Metacarpophalangeal joint mechanics after 3 different silicone arthroplasties. J Hand Surg Am. 2004 Sep;29(5):796-803. doi: 10.1016/j.jhsa.2004.04.023. PMID 15465227